CLINICAL TRIAL: NCT00055380
Title: Molecular, Genetic, and Biochemical Effects Of Novel Therapies In Buccal Mucosal Cells
Brief Title: Chemical and Genetic Effects of the Experimental Anti-Cancer Drugs in Cheek Cells in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030115; 03-D-0115
Record Dates: First submitted 2003-02-28; First posted 2003-02-28 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Cancer
Keywords: Molecular Targets; Keratinocytes; Cell Cycle; Small Molecule; Gene Expression; Pharmacodynamics; Surrogate Markers; Targeted Therapy; Buccal Mucosa; Pharmacogenomics; Oral Mucosa
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Procedure: Oral cytobrushing

SUMMARY:
This study will examine the effects of certain investigational anti-cancer drugs on the genetic and protein makeup of cells. The findings will be entered into a database that may be used to: 1) determine the optimal dose of drug that will provide the most benefit with the least harmful side effects; and 2) predict which patients will have a greater chance of developing side effects or a greater chance of benefiting from the drug.

Patients 18 years of age and older who are receiving the anti-cancer drugs flavopiridol or perifosine in an NIH clinical trial may be eligible for this study.

Participants will undergo the following procedures both before starting treatment and during the first treatment cycle to look for genetic or chemical changes produced in response to the study drug:

* Blood draws.
* Buccal cell brushings: Collection of buccal cells (cells lining the inside of the cheeks) from the inside of the cheeks using a soft bristle brush for a few seconds several times. The patient then rinses the mouth with salt water for 1 minute and then spits into a cup.
* Buccal cell biopsies (on both sides of the mouth): For this procedure, a local anesthetic is given to numb the biopsy area. Then, a small piece of tissue from the inner lining of the mouth is removed with a small sharp cookie-cutter instrument. The biopsy findings will be compared with those of the cheek brushings to see if the information is similar.
* Tumor biopsies: In patients whose tumor is easily accessible, such as the skin abdominal fluid, tissue biopsies will be requested. Depending on the type and location of the tumor, the biopsy may be done with a forceps, a large needle (needle biopsy), a cookie-cutter instrument (punch biopsy), or a small knife (excisional biopsy). All of these procedures are done with a local anesthetic.

DETAILED DESCRIPTION:
A significant problem in drug development of novel small molecules is the lack of available tissues (surrogate tissues) that allow for the assessment of the molecular and biochemical effects of (targeted-therapies) drug action. The information obtained from surrogate tissues might help us validate previous preclinical studies with those agents and also dose them in a more rational way. Oral keratinocytes, which are accessible by non-invasive means, might be useful to assess drug action. The proposed study seeks to investigate the genetic, molecular, and biochemical effects of novel agents in oral buccal mucosal cells. Patients already enrolled in Phase I and II clinical trials for neoplastic diseases at the Clinical Center will undergo oral cytobrushing before and during therapy to determine the molecular and biochemical effects of novel agents in the oral mucosa cells. Similar studies will be performed in peripheral blood mononuclear cells. In order to validate to compare and compare the oral cytobrush methodology, some of these subjects will undergo oral punch biopsy studies. Some of these subjects will also undergo tumor biopsy, if accessible or available.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients (male, female, greater than or equal to age 18 years) enrolled in a clinical trial at the Clinical Center receiving novel small molecules that modulate cell cycle progression for the prevention and treatment of neoplastic diseases.

Able to sign informed consent.

Patient's primary NIH physician should agree with appropriateness of patient's participation in the study.

EXCLUSION CRITERIA:

Patients unable to undergo cytobrushing (significant mucositis).

Non-compliant patients.

Patients unable to provide baseline samples (patients already receiving therapy).

Exclusion for biopsy only: patients with significant bleeding diathesis, receiving active anticoagulation or with platelets less than 10K.

Cognitively impaired subjects will be excluded from this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2003-02; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Senderowicz AM. Small molecule modulators of cyclin-dependent kinases for cancer therapy. Oncogene. 2000 Dec 27;19(56):6600-6. doi: 10.1038/sj.onc.1204085. PMID 11426645
- [Background] Senderowicz AM, Sausville EA. Preclinical and clinical development of cyclin-dependent kinase modulators. J Natl Cancer Inst. 2000 Mar 1;92(5):376-87. doi: 10.1093/jnci/92.5.376. PMID 10699068
- [Background] Buolamwini JK. Cell cycle molecular targets in novel anticancer drug discovery. Curr Pharm Des. 2000 Mar;6(4):379-92. doi: 10.2174/1381612003400948. PMID 10788588